CLINICAL TRIAL: NCT06618170
Title: Evaluation Clinique Des Performances Du Dispositif D'Aide À La Chirurgie Dyameo
Acronym: ETCETERA
Status: Not yet recruiting | Type: Observational
Sponsor: Dyameo (Industry)
Collaborators: GETTEC (Groupe d'Etude des Tumeurs de la Tête et du Cou) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A01462-45
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Cancers
Keywords: guided surgery; head and neck; carcinoma; surgical margin
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma; Margins of Excision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Tissue surface analysis with the device — Usage of the device to analyse the presence or absence of tumoral membrane marker at the surface of the removed tumoral specimen

SUMMARY:
During the surgical removal of head and neck tumours, the correct determination of the boundary between healthy and tumour tissue is critical. It is essential to remove all tumour tissue while preserving as much of the surrounding healthy tissue as possible. Today, surgeons use frozen sections to confirm their decision. Dyameo has developed a device that can identify the presence of tumour markers on the surface of tissue in a matter of seconds, simply by placing the end of a fibre-optic probe in contact with the tissue. This device should enable the surgeon to identify the presence of tumour cells at the margin of the removed tumour.

The aim of this study is to measure the performance of this device. The surgeon will carry out his operation according to his own routine. After collecting tissue for frozen section analysis, he will analyse the tumour specimen using the Dyameo device. After the operation, histological analysis of the removed tumour will enable the precision of the device to be measured and compared with that of the extemporaneous biopsies to guide the surgeon's intervention.

DETAILED DESCRIPTION:
This will be a mThe surgeon will remove the tumour and collect frozen section according to his usual practices. He will then analyse the same areas on the specimen, or directly analyse the tissue sampled for the frozen section using the Dyameo device. The position of the analysis will be marked on the specimen by sutures. No results will be displayed on the screen at this stage, so as not to influence the doctor;s actions. The surgeon is also free to analyse additional areas with Dyameo device if he or she considers this to be of interest. After the operation, the pathology lab will analyze the tumor specimen to assess the margin status and evaluate the exact nature of the tissues on the localisation of frozen section/Dyameo analysis. Simultaneously, the results of the analyses carried out with the Dyameo device will be exported and analysed (blind to the results of the histological analysis), in order to determine the indications that would have been given to the surgeon during the operation.

The results obtained with the device will be compared with the results of the extemporaneous biopsy analysis. The postoperative histological analysis will serve as a reference.

The performance of the device will be measured by evaluating a posteriori the accuracy of the results provided, and therefore the accuracy of the instructions given to the surgeon during the operation (e.g. additional recutting in the event of the presence of residual tumour cells at the margin of the tumour specimen). The study will also make it possible to calculate sensitivity, specificity, precision, positive and negative predictive values, and relative risk for the device.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of squamous cell carcinoma of the oral cavity, pharynx and/or larynx
* Planned standard surgery with curative intent for squamous cell carcinoma
* Planned surgery includes the performance of extemporaneous biopsies
* Age ≥ 18 years
* Affiliation to a social security scheme

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to understand the research in which he or she is participating
* Persons of full age subject to a legal protection measure (guardianship or curatorship) or unable to express their non-objection.
* Uncontrolled concomitant medical conditions
* Having received an investigational medicinal product in the 30 days prior to the operation
* History of treatment with anti-EGFR monoclonal antibodies.
* Previously demonstrated absence of EGFR expression by tumour cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with squamous cell carcinoma of head and neck for whom surgical removal requiring frozen section analysis is planned.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Dyameo device in guiding surgical procedures | During the surgical intervention
  Proportion of cases where analysis with the Dyameo device has provided valid instructions to guide surgery (e.g. make an additional cut if tumour cells are present in at least one area of the resection margin)

SECONDARY OUTCOMES:
Device performances | During the surgical intervention
  Sensibility, specificity, positive and negative predictive value, relative risk of the device

IPD SHARING:
Plan to Share IPD: Undecided